CLINICAL TRIAL: NCT06254001
Title: Effectiveness of Combined Treatment of Bupropion and Nicotine Replacement Therapy in Hospitalized Subjects With Active Smoking in a Reference Center
Brief Title: Effectiveness of Combined Tobacco Treatment in Hospitalized Subjects
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Ireri Thirion Romero, Principal Investigator, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C80-23
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Smoking; Tobacco Withdrawal; Nicotine Addiction; Nicotine Withdrawal; Nicotine Replacement Therapy
Keywords: tobacco; bupropion; nicotine replacement therapy; abstinence
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use Disorder | interventions — Bupropion; Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Two groups:
  1. Nicotine replacement therapy
  2. Nicotine replacement therapy and bupropion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine replacement therapy (Active Comparator): Nicotine replacement therapy (Nicotine patches) plus counseling and cognitive behavioral therapy
  Interventions: Drug: Nicotine replacement therapy (Nicotine patches)
- Nicotine replacement therapy and Bupropion (Experimental): Nicotine replacement therapy (Nicotine patches) plus Bupropion and counseling and cognitive behavioral therapy
  Interventions: Drug: Bupropion; Drug: Nicotine replacement therapy (Nicotine patches)

INTERVENTIONS:
Drug: Bupropion — Bupropion will be added at doses of 150 mg to 300 mg per day in addition to nicotine replacement therapy, counseling and cognitive behavioral therapy
  Arms: Nicotine replacement therapy and Bupropion
Drug: Nicotine replacement therapy (Nicotine patches) — Nicotine replacement therapy (Nicotine patches) plus counseling and cognitive behavioral therapy

SUMMARY:
In the 20th century, tobacco caused the death of 100 million people worldwide and it is estimated that it will be responsible for 1 billion deaths in the 21st century. Currently 8 million people die each year from smoking, 7 million are associated with active smoking, thus being the main risk factor for loss of disability-adjusted life years for men and the ninth most important risk factor for women. In previous studies it has been reported that approximately 21% (14%-30%) of subjects who have required hospitalization are active smokers, being higher in men than in women (28% vs 14%). The initiation of treatment for smoking cessation in this group of subjects has shown an effectiveness rate of up to 65% to maintain abstinence 6 to 12 months after discharge. The effectiveness has been analyzed in scenarios with only brief advice, in some others with the use of medications such as varenicline, bupropion and nicotine replacement therapy, however, the interventions have not been standardized for adequate analysis, which could contribute to the different results.

DETAILED DESCRIPTION:
The objective is to know the effectiveness of combined treatment to maintain abstinence in participants with active smoking who are hospitalized in a reference center.

Bupropion and nicotine replacement therapy are the drugs used in this clinical trial.

Participants will be randomly assigned to two groups: nicotine replacement therapy or nicotine replacement therapy plus bupropion. All participants will have counseling, conductive behavioral therapy, follow-up at 3, 6 and 12 months with a pulmonologist. Pulmonary function tests will be performed every 3, 6, and 12 months. Abstinence will be corroborated with a cotinine (urine) test and an exhaled carbon monoxide test.

ELIGIBILITY:
Inclusion Criteria:

>18 years Active smokers (consumption of more than 100 cigarettes in their entire life, and who have consumed cigarettes in the last 30 days) Hospitalized subjects Informed consent

Exclusion Criteria:

* Subjects who have had pharmacological treatment to stop smoking in the last month
* Subjects with contraindications for medications.

Sample size calculation, 80% power, unilateral, due to difference in proportions, estimated loss of 25%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Abstinence at 12 months. Negative cotinine test and negative an exhaled carbon monoxide test | 12 months
  Abstinence will be corroborated with a cotinine test and an exhaled carbon monoxide test. Negative urine cotinine test and an exhaled carbon monoxide test less than 6 ppb.

CONTACTS AND LOCATIONS:
Overall Officials: IRERI THIRION-ROMERO, DR, Principal Investigator — INER
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data will be collected on the redCap platform, and may be shared in Excel CSV format as well as related dictionaries. SAP, ICF, CSR information will be shared after the results are published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD data will be available when the study is published in December 2026 and will remain for an additional year until December 2027.
Access Criteria: The information may be requested by researchers who wish to carry out meta-analysis or researchers related to the area of secondary prevention of smoking. They may request it from the main or corresponding author who will review the applications.

REFERENCES:
- [Background] Martinez C, Fu M, Castellano Y, Riccobene A, Fernandez P, Cabrera S, Gavilan E, Feliu A, Puig-Llobet M, Fuster P, Martinez-Sanchez JM, Montes J, Estrada JM, Moreno C, Falco-Pegueroles A, Galimany J, Brando C, Suner-Soler R, Capsada A, Fernandez E; y Grupo de Coordinadores de la Red Catalana de Hospitales sin Humo (XCHsF). Smoking among hospitalized patients: A multi-hospital cross-sectional study of a widely neglected problem. Tob Induc Dis. 2018 Jul 30;16:34. doi: 10.18332/tid/92927. eCollection 2018. PMID 31516433
- [Background] Rigotti NA, Clair C, Munafo MR, Stead LF. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2012 May 16;5(5):CD001837. doi: 10.1002/14651858.CD001837.pub3. PMID 22592676
- [Result] Makate M, Whetton S, Tait RJ, Dey T, Scollo M, Banks E, Norman R, Pidd K, Roche AM, Allsop S. Tobacco Cost of Illness Studies: A Systematic Review. Nicotine Tob Res. 2020 Apr 17;22(4):458-465. doi: 10.1093/ntr/ntz038. PMID 30874290
- See also: Tobacco Control is an international peer-reviewed journal covering the nature and consequences of tobacco use worldwide — https://tobaccocontrol.bmj.com/?utm_source=google&utm_medium=search&utm_campaign=usage&utm_term=usage&gclid=Cj0KCQiAn-2tBhDVARIsAGmStVn8-mzKFk9rRlFCYB6-4QNsMKYq4FGv6-5sFxHl-NENwHwJO8GlsbQaAlnREALw_wcB

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT06254001/Prot_SAP_000.pdf